CLINICAL TRIAL: NCT06355661
Title: A Double-blind, Randomized, Placebo-Controlled, Comparative Study for Assessing the Efficacy and Safety of ParActin® in Individuals With Upper Respiratory Tract Infections (URTI)
Brief Title: A Study for Assessing the Efficacy and Safety ParActin® in Individuals With Upper Respiratory Tract Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP/231102/PA/URTI
Record Dates: First submitted 2024-03-21; First posted 2024-04-09 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-03

CONDITIONS: Upper Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: A Double-blind, Randomized, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ParActin®: 300 mg + MCC: 100 mg (± 10%) (Active Comparator): Two capsules/day (One capsule to be taken 30 minutes before breakfast & one capsule to be taken 30 minutes before dinner).
  Interventions: Dietary Supplement: ParActin®: 300 mg + MCC: 100 mg (± 10%) per Capsule
- MCC: 400 mg (± 10%) per Capsule (Placebo Comparator): Two capsules/day (One capsule to be taken 30 minutes before breakfast & one capsule to be taken 30 minutes before dinner).
  Interventions: Dietary Supplement: MCC: 400 mg (± 10%) per Capsule

INTERVENTIONS:
Dietary Supplement: ParActin®: 300 mg + MCC: 100 mg (± 10%) per Capsule — Two capsules/day (One capsule to be taken 30 minutes before breakfast & one capsule to be taken 30 minutes before dinner)
  Arms: ParActin®: 300 mg + MCC: 100 mg (± 10%)
Dietary Supplement: MCC: 400 mg (± 10%) per Capsule — Two capsules/day (One capsule to be taken 30 minutes before breakfast & one capsule to be taken 30 minutes before dinner)
  Arms: MCC: 400 mg (± 10%) per Capsule

SUMMARY:
The present study is a randomized, double-blind, placebo-controlled, comparative study. 176 individuals will be screened, and considering a screening failure rate of 15 percent approximately 150 will be randomized in a ratio of 1:1 to receive either IP or placebo and will be assigned a unique randomization code. Each group will have at least 60 completed participants after accounting for a dropout/withdrawal rate of 20percent. The intervention duration for all the study participants is 7 days

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged between 18 and 50 years as of the screening date.
2. Individuals with symptoms of acute upper respiratory tract infection as assessed by the investigator at the time of screening.
3. BMI ≤ 29.9 kg/m2.
4. Upper respiratory tract infection symptoms present for at least 24 hours but not more than 48 hours prior to screening visit.
5. Those having a score of ≥ 5 for at least 2 symptoms out of runny nose, plugged nose, sneezing or sore throat, on the WURSS-21.
6. History of frequent common cold with past episode duration of at least 4 days.
7. Must be literate and have the ability to complete the study-based questionnaires and requirements.

Exclusion Criteria:

1. High grade fever defined as body temperature ≥ 39ºC (≥ 102.2 ºF)
2. With a history of allergy (allergic rhinitis) along with symptoms such as sneezing, runny nose and red, watery and itchy eyes.
3. Individuals with history of Chronic obstructive pulmonary disease, pulmonary fibrosis or Asthma.
4. Individuals with rhinitis medicamentosa, chronic cough of bacterial, fungal or other known origin.
5. Individuals requiring hospitalization or likely to be hospitalised due to URTI.
6. Individuals with common cold for the first time.
7. Individuals with anatomical nasal obstruction/ deformity or nasal reconstructive surgery etc.
8. Individuals with history of heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies
9. Individuals with history of immunocompromised state immune system with/ without organ transplant
10. Individuals with known or suspected hypersensitivity or intolerance to herbal products
11. Individuals diagnosed with Sickle cell disease, Thalassemia, Type I/ II Diabetes mellitus, Cystic fibrosis
12. Diagnosed cases of Uncontrolled hypertension as assessed by a systolic blood pressure ≥ to 140mmHg and diastolic blood pressure ≥ to 90mmHg
13. Those not willing to abstain from home based cold remedies that include but are not limited to steam inhalation, decoctions, vapour rub, ginger supplement, decoctions, or any form of dietary and/or herbal supplements during the entirety of study participation period.
14. Those who have been vaccinated for influenza, swine flu 3 months prior to screening visit.
15. Those who have taken within one week of the start of the study or require during study antibiotics, antivirals, steroids, nasal decongestants, antihistamines herbal remedies, Vitamin C or Zinc to alleviate cold symptoms.
16. Those who have severe mental illnesses, such as dementia, Parkinson's disease, Alzheimer's Disease, depression or anxiety disorders, or those who are currently taking psychoneurological drugs, such as antidepressants.
17. Those who have participated in other clinical study within 30 days, prior to the screening visit or plan to participate in other clinical study during the study period.
18. Individuals with substance abuse as per last two-year history that includes the use of but is not limited to drugs such as cocaine, amphetamine, marijuana etc.
19. Individuals having a history of smoking or currently smoking or using any form of smokeless tobacco.
20. Individuals with heavy alcohol consumption, defined as:

    1. For men: More than 14 standard alcoholic drink (SAD)/week or more than 4 SAD in a day.
    2. For women: More than 7 SAD/week or more than 3 SAD in a day.
    3. Binge drinkers, defined as 5 or more SAD for men, in a 2-hour time frame.
    4. Binge drinkers, defined as 4 or more SAD for Women, in a 2-hour time frame. (NOTE - A standard alcoholic drink contains approximately 14 grams of alcohol, which is equivalent to 12 ounces of beer (~5% alcohol), 8.5 ounces of malt liquor (~9% alcohol), 5 ounces of wine (~12% alcohol), 3.5 ounces of fortified wine (e.g., sherry or port), or 1.5 ounces of liquor (distilled spirits; ~40% alcohol)
21. Those who have clinically significant disorder/s of cardiovascular, endocrine, lymphatic, respiratory, hepatobiliary, urinary, reproductive, central nervous system, musculoskeletal and digestive systems.
22. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
23. Any condition that could, in the opinion of the investigator, preclude the individual's ability to successfully and safely complete the study or that may confound study outcomes.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of investigational products on participant's severity of common cold like symptoms | During Upper respiratory tract infection episodes throughout the study upto 7 day Treatment duration
  evaluated by Wisconsin Upper Respiratory Symptom Survey-21 total severity score (incremental Area Under the Curve (iAUC) The WURSS-21 consists of ten symptom-specific items which includes runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion, and feeling tired.

SECONDARY OUTCOMES:
To evaluate the effect of investigational products on Time (in days) taken to resolution of common cold like symptoms | During episodes of URTI upto 7 day Treatment duration
  resolution deemed to occur when participant reports being "0 = not sick" as per Wisconsin Upper Respiratory Symptom Survey-21 for two consecutive days during the treatment period, The WURSS-21 consists of ten symptom-specific items which includes runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion, and feeling tired.
To evaluate the effect of investigational products on Percentage of participants with unresolved common cold symptoms | During episodes of URTI upto 7 day Treatment duration
  being those who do not report being "0 = not sick" as per Wisconsin Upper Respiratory Symptom Survey-21 till the end of the treatment period.
  An episode is deemed resolved when the participant marks "0 = not sick" on Q.1 of WURSS-21 for two consecutive days. If this criterion is not met, the episode is considered unresolved
To evaluate the effect of investigational products on Percentage of population with minimal important difference of ≥ 10.3 as per change in Wisconsin Upper Respiratory Symptom Survey-21 total score. (daily score will be analysed in study) | During episodes of URTI upto 7 day Treatment duration
  The WURSS-21 consists of ten symptom-specific items which includes runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion, and feeling tired
To evaluate the effect of investigational products on Number of days taken to be afebrile (temp < 100 oF/< 37.7 ºC) in the population with fever (temp ≥100oF or ≥37.7 ºC ) at baseline- as assessed by 10-point visual analogue scale. | During episodes of URTI upto 7 day Treatment duration
  Place the thermometer in the armpit. Press the arm against the body. Wait for 2-3 minutes before reading in case of traditional thermometer or until it beeps in case of digital thermometer. The number of days taken to be afebrile (temp < 100 oF or < 37.7 ºC) in the population with fever (temp ≥100oF or ≥37.7 ºC ) at baseline will be recorded. The participants will record their fever daily on diary
To evaluate the effect of investigational products on Percentage population with fever during the study. | During episodes of URTI upto 7 day Treatment duration
  Place the thermometer in the armpit. Press the arm against the body. Wait for 2-3 minutes before reading in case of traditional thermometer or until it beeps in case of digital thermometer. The number of days taken to be afebrile
To evaluate the effect of investigational products on Quality of life as assessed by Wisconsin Upper Respiratory Symptom Survey Quality of Life | Day 0, day 4 and day 8
  The Wisconsin Upper Respiratory Symptom Survey-21 consists of ten symptom-specific items which includes runny nose, plugged nose, sneezing, sore throat, scratchy throat, cough, hoarseness, head congestion, chest congestion, and feeling tired.All the items will be scored on an 8-point Likert scale ranging from 0 which depicts "absent or no impairment" through 1 (very mild), 3 (mild), 5 (moderate) and 7 (severe)

CONTACTS AND LOCATIONS:
Locations (9):
- India (9):
  - Life care hospital, Nashik, Maharashtra
  - ENT Vertigo Clinic, Pune, Maharashtra
  - Jawaharlal Nehru Medical College, Ajmer, Rajasthan
  - Human Care Hospital, Lucknow, Uttar Pradesh
  - Shubham Sudbhawana Super Speciality Hospital, Varanasi, Uttar Pradesh
  - Janta Hospital, Varanasi, Uttar Pradesh
  - Gastron Clinic, Delhi
  - Good health Clinic, Delhi
  - Tulsi Multispecility Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No